CLINICAL TRIAL: NCT01868984
Title: The Use of Intravascular Paclitaxel for the Treatment of Upper-Extremity Arteriovenous Access Fistula Stenosis: A Randomized Study
Brief Title: Paclitaxel for the Treatment of Upper-Extremity Arteriovenous Access Fistula Stenosis
Acronym: PaciFIST-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: catheters no longer available - difficult to recruit subjects
Sponsor: Englewood Hospital and Medical Center (Other)
Collaborators: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-12-468
Record Dates: First submitted 2013-05-29; First posted 2013-06-05 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Fistula Stenosis
MeSH Terms: interventions — Paclitaxel; Standard of Care; Heparin; Stents; Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy Alone (Sham Comparator): Standard treatment of all stenotic lesions will be carried out in the usual fashion. Intravenous heparin will be administered in a standard dose of 70 units/kg. Lesions that respond poorly to angioplasty (>30% residual stenosis after angioplasty treatment with 2 inflations) will be stented. Stent selection will be based on clinical setting. Initial stent treatment will utilize an uncovered nitinol stent. Treatment of in-stent restenosis will include initial balloon angioplasty, and use of a covered stent (Viabahn, GORE, or Fluency, Bard).
  For this "control" group, no paclitaxel is administered. The sham treatment is a period of 10 minutes that is allowed to elapse followed by the performance of a final completion angiogram to be labeled as "PaciFIST Study Completion Angiogram." Any additional lesions identified with this study are then treated appropriately following standard technique.
  Interventions: Procedure: Standard Therapy
- Standard Therapy Plus Paclitaxel (Active Comparator): Standard treatment of all stenotic lesions will be carried out in the usual fashion. Intravenous heparin will be administered in a standard dose of 70 units/kg. Lesions that respond poorly to angioplasty (>30% residual stenosis after angioplasty treatment with 2 inflations) will be stented. Stent selection will be based on clinical setting. Initial stent treatment will utilize an uncovered nitinol stent. Treatment of in-stent restenosis will include initial balloon angioplasty, and use of a covered stent (Viabahn, GORE, or Fluency, Bard).
  For this "treatment" group, Paclitaxel solution treatment of each lesion encountered from proximal to distal will be attempted until the 20 mg Paclitaxel dose limit is met.
  Interventions: Drug: Paclitaxel; Procedure: Standard Therapy

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel solution treatment of each lesion encountered will be attempted until the 20 mg Paclitaxel dose limit is met. The volume administered will depend on the diameter and length of the venous outflow segment.
  Other Names: Taxol
  Arms: Standard Therapy Plus Paclitaxel
Procedure: Standard Therapy — Standard treatment of all stenotic lesions will be carried out in the usual fashion. Intravenous heparin will be administered in a standard dose of 70 units/kg. Lesions that respond poorly to angioplasty (>30% residual stenosis after angioplasty treatment with 2 inflations) will be stented. Stent selection will be based on clinical setting. Initial stent treatment will utilize an uncovered nitinol stent. Treatment of in-stent restenosis will include initial balloon angioplasty, and use of a covered stent (Viabahn, GORE, or Fluency, Bard).
  Other Names: heparin; stents; angioplasty

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the use of intravascular paclitaxel, in addition to standard therapy, for the treatment of arteriovenous dialysis access fistula stenosis.

A fistulogram will be performed in standard fashion. The diagnostic component will include evaluation of the inflow artery, arterial anastomosis and full length of the fistula vein or graft, plus venous return up to the heart. The location, vessel size, lesion diameter and percent stenosis for each lesion will be recorded. Enrollment and randomization will occur at this point.

All patients will then receive standard therapy for their stenosis. This will include intravenous heparin administered in a standard dose of 70 units/kg. Lesions that respond poorly to angioplasty (>30% residual stenosis after angioplasty treatment with 2 inflations) will be stented. Stent selection will be based on clinical setting. Initial stent treatment will utilize an uncovered nitinol stent. Treatment of in-stent restenosis will include initial balloon angioplasty, and use of a covered stent (Viabahn, GORE, or Fluency, Bard). Documentation of location and type of treatment for each lesion treated will be recorded.

Once standard treatment is completed, the operating surgeon will be informed of the patient randomization: treatment (paclitaxel) or control. For subjects assigned to treatment, Paclitaxel solution treatment of each lesion encountered from proximal to distal will be attempted until the 20 mg Paclitaxel dose limit is met.

A TAPAS infusion catheter will be used for all paclitaxel dose administrations. The TAPAS infusion catheter will be positioned to reduce the presence of branches which permit the loss of paclitaxel from the treatment zone. After the full outflow vein segment is treated, the fistulogram is completed in the standard fashion. Prior to removal of the sheath, a final angiographic study of all areas treated is performed to document patency and lesion appearance.

For the control group, instead of paclitaxel administration, a sham treatment period of 10 minutes is allowed to elapse followed by the performance of the final completion angiogram. Any additional lesions identified with this study are then treated appropriately following standard technique.

All patients will follow the same follow up evaluation schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patient or guardian able to provide a signed witnessed informed consent
3. Stenosis greater than or equal to 50% treated satisfactorily (less than 20% residual stenosis) with balloon angioplasty alone or balloon angioplasty and stent placement
4. Either gender

Exclusion Criteria:

1. Women who are pregnant or who are expected to or might become pregnant
2. Women of child-bearing potential who do not use contraception
3. Life expectancy less than 12 months
4. Known allergy to paclitaxel
5. Known allergy to contrast media not previously demonstrated to be controllable with premedication on a prior study using contrast
6. Known allergy to the pre-medications (dexamethasone, famotidine, diphenhydramine)
7. Pre-fistulogram thrombosis of the fistula or graft
8. Thrombectomy of the fistula or graft within 14 days of the procedure
9. Patient receiving chemotherapy
10. Patients with an immunodeficiency disease or condition
11. Documented hypercoagulable state
12. White Blood Count < 2000/mm3
13. Platelet count less than 100,000/mm3
14. Chronic hepatitis or jaundice (total bilirubin > 2x upper limit of normal)
15. Simultaneous enrollment in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Target Lesion Revascularization. | 6 months
  Target lesion revascularization (TLR) is defined as the need for subsequent clinically driven repeat angioplasty, stent placement or other intervention to correct the recurrence of a stenosis at the site treated within 6 months of the initial treatment.
Target Segment Revascularization. | 6 months
  Target segment revascularization (TSR) is defined as the need for secondary clinically driven repeat angioplasty, stent placement or other intervention to correct the recurrence of a stenosis in the outflow segment of cephalic vein treated with paclitaxel.

SECONDARY OUTCOMES:
Overall safety based on SAEs | 6 months
  The overall serious adverse event (SAE) rate will be determined as well as the rate for each individual type of adverse occurrence or event.
Binary Restenosis | 6 months
  The development of recurrent stenosis of the site treated with angioplasty or angioplasty and stent followed by the paclitaxel controlled infusion. The presence of a binary stenosis is defined as a 50% decrease of the vessel diameter measured on the fistulogram.
Primary Patency: Fistula | 6 months
  The interval from treatment until access thrombosis or repeat intervention treatment to maintain fistula function, or the abandonment of the fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Wengerter, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States

REFERENCES:
- See also: Related Info — https://www.englewoodhealth.org/service/clinical-research-center/open-clinical-trials